CLINICAL TRIAL: NCT03337230
Title: A Pilot Intervention Study to Examine the Feasibility of a Social Media-Based Weight Loss Program for Low Socioeconomic Status Individuals
Brief Title: Feasibility of a Social Media-based Weight Loss Program for Low Socioeconomic Status Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CASE17Z17
Record Dates: First submitted 2017-11-06; First posted 2017-11-08 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Obesity
Keywords: Cancer; Weight-Loss; Social Media
MeSH Terms: conditions — Obesity; Neoplasms; Weight Loss | interventions — Exercise; Diet

STUDY DESIGN:
Intervention Model Description: pre-post study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity + Diet + Social media (Experimental): Educational materials for the proposed study will be delivered via a secret social media Facebook group. These materials will promote simple, attainable forms of Physical Activity and lasting diet changes. A study moderator will deliver weekly communications to the Facebook group providing intervention content including social support, social competition and comparison, and social rewards
  Interventions: Behavioral: Physical Activity; Behavioral: Diet; Behavioral: Social Support

INTERVENTIONS:
Behavioral: Physical Activity — Fitbit Activity Monitor and IPAQ to give level of physical activity. Participants will be provided with education about physical activity recommendations and will be encouraged to set goals for improvement.
Behavioral: Diet — National Cancer Institute's ASA24 web-based dietary assessment tool to determine intake. Participants will be provided with education about healthy diets and will be encouraged to set goals for making enduring changes to dietary intake.
Behavioral: Social Support — Social support will be determined via self report scale measure and objective collection of social media communications. Each participant will be contacted through social media regularly with dietary and physical activity information and asked to support other participants via encouragement and sharing of information.

SUMMARY:
The purpose of this study is to see if it is practical to use social media-based and traditional online weight loss intervention components among low socioeconomic status participants using the Facebook social media (SM) and Fitbit self-monitoring platforms. Also, the study will test the effectiveness of recruiting participants via social media and at community events and locations. The results of this study will be used to inform future research studies.

DETAILED DESCRIPTION:
The primary objectives of the proposed research are to:

1. assess the feasibility of social media-based (social support, social competition, and social rewards) and traditional online weight loss (education and goal setting) intervention components delivered to low-Socioeconomic Status (SES) participants using the Facebook SM and Fitbit self-monitoring platforms and
2. develop and assess methods for recruiting and retaining adequate numbers of low-SES participants for a future randomized controlled trial to assess the efficacy of an SM-based weight loss intervention. The study team will assess feasibility by conducting a 12-week pilot test of traditional and social media-based weight loss intervention components followed by qualitative and quantitative assessment with pilot participants.

The specific aims are:

Aim 1- Assess trial feasibility: The study team will assess intervention processes critical to the success of a larger efficacy trial during the 12-week pilot including: (1) participant recruitment and retention, (2) participant use of intervention components, (3) use of data collection strategies and instruments.

Aim 2 - Assess intervention acceptability: The study team will conduct structured interviews and surveys among participants to assess participants' experience during the intervention. This study focuses on: (1) intervention design and content, (2) participant use of intervention technologies (Facebook and Fitbit), (3) participant concerns about privacy, and (4) barriers and facilitators to recruitment, retention, and participation. Findings will be used to improve the design of a larger efficacy trial.

Study Design: This study will employ a one group pre-post design.

ELIGIBILITY:
Inclusion Criteria:

* able to speak English
* regular access to an internet-enabled device that can be synched with the Fitbit wristband
* Body mass index (BMI) 25-40 kg/m^2
* < 30 minutes per day of self-reported moderate or vigorous physical activity
* Considered eligible for Ohio Expanded Food and Nutrition Education Program (EFNEP) income guidelines
* located in the greater Cleveland metropolitan area
* not pregnant or planning on becoming pregnant
* answers 'no' to all questions on the PA Readiness Questionnaire (PAR-Q) or is cleared in writing by a physician
* does not have a recent history of alcohol or drug abuse or is in treatment
* does not have schizophrenia

Exclusion Criteria:

* Does not meet all inclusion criteria

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Ratio or participants screened to patients completing 12-week measures | Up to 12 weeks
  This is a measure of feasibility
Average score of adapted INSHAPE computer-based questionnaire | Up to 12 weeks
  Computer-based questionnaires will be self-administered via the Qualtrics Survey platform. INSHAPE questionnaire is a 14 question survey gauging acceptability of the program

SECONDARY OUTCOMES:
Number of eligible participants | Up to 12 weeks
  This is a measure of feasibility
Number of consented participants | Up to 12 weeks
  This is a measure of feasibility
Average change in Fitbit activity | From baseline to 12 weeks
  This is a measure of physical activity
Average change in International physical activity questionnaire (IPAQ) score | From baseline to 12 weeks
  This is a measure of physical activity
Average change in score of the National Cancer Institute's Automated Self-Administered 24-Hour (ASA24) dietary assessment web-based assessment tool | From baseline to 12 weeks
  This is a measure of dietary intake
Change in weight | From baseline to 12 weeks
  Trained study staff will determine weight at baseline and 12 weeks of the study
Change in waist circumference | From baseline to 12 weeks
  Trained study staff will determine waist circumference at baseline and 12 weeks of the study
Average change in social support score | From baseline to 12 weeks
  This is a 31 question, multiple choice survey adapted from Gruber and Sallis
Average change in weight loss self-efficacy score | From baseline to 12 weeks
  Multiple choice questions and short answer survey which can be scored to gauge weight-loss self-efficacy. Adapted from Wilson
Average change in dietary knowledge | From baseline to 12 weeks
  Multiple choice questions and short answer survey which can be scored to gauge dietary knowledge. Adapted from Jones

CONTACTS AND LOCATIONS:
Overall Officials: David N. Cavallo, PhD MPH RDN, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Western Reserve Univeristy, Cleveland, Ohio, United States